CLINICAL TRIAL: NCT01416532
Title: Prognostic Value of Coronary CT Angiography in Relation to Evaluation of Subclinical Coronary Atherosclerosis for Risk Stratification in Asymptomatic Individuals From ESCORT Study
Brief Title: Evaluation of Subclinical COronary Atherosclerosis for Risk Stratification Using Coronary Computed Tomography (CT) Angiography
Acronym: ESCORT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Seoul National University Bundang Hospital, Seoul National University Bundang Hospital
Other Study IDs: B-1107-131-104
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Atherosclerosis
Keywords: coronary Atheroslcerosis; Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To evaluate the prognostic value of coronary CT angiography (CCTA) for risk stratification in asymptomatic adults in comparison with conventional risk stratification (CRS) and coronary artery calcium scoring (CACS).

DETAILED DESCRIPTION:
The risk stratification of cardiovascular disease (CVD) in asymptomatic individuals represents a major challenge. For this purpose, a lot of risk prediction models that take demographic and clinical characteristics into account have been developed. Although Framingham risk score (FRS) is most widely used among multiplr risk prediction models, it has some limitation for prediction of CVD especially in young adult and women. Recently, coronary artery calcium score (CACS) has known to be powerful screening method for CVD, however, it cannot detect the noncalcified coronary plaques (NCP), so it does not represent the entire spectrum of atherosclerotic plaques and it also cannot evaluate the degree of stenosis. On the contrary, Coronary CT angiography (CCTA)can provide detailed coronary artery anatomy and plaque imaging about the location, burden and characteristics of atherosclerotic plaque per se, which might give additional insight to stratify the risk of future cardiac events and therapy.

In this study, we will evaluate the prevalence and characteristics of subclinical coronary atherosclerosis on CCTA in asymptomatic population. And we will investiage the follow up data for major cardiac adverse event such as cardiac death, nonfatal myocardial infarction, unstable angina and revascularization. Therefore, we will finally evaluate the prognostic value of CCTA for risk stratification in asymptomatic adults in comparsion with conventional risk stratification such as FRS and CACS.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic subjects
* adults > 20 years
* subjects who underwent both calcium score and coronary CT angiography

Exclusion Criteria:

* typical or atypical chest pain
* subjects who underwent previous percutaneous coronary intervention
* serious comorbid conditions(i.e. malignancy)
* insufficient medical record
* poor image quality

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymptomatic adults without previous coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eun Ju Chun, MD, PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seound National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Yoo JY, Kang SR, Bae YJ, Chun EJ. Comparison of Cardiac Events and Survival Between Asymptomatic Diabetic and Nondiabetic Patients: Coronary CT Study. J Korean Med Sci. 2025 Oct 20;40(40):e251. doi: 10.3346/jkms.2025.40.e251. PMID 41120106